CLINICAL TRIAL: NCT01654276
Title: Effects of Pharmacological Reversal of Hyperuricemia on Features of the Metabolic Syndrome
Brief Title: Effects of Hyperuricemia Reversal on Features of the Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Naim Maalouf, Assistant Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSA-FEB-137
Record Dates: First submitted 2012-06-28; First posted 2012-07-31 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Febuxostat (Experimental): Adult patients (age > 21 years) with gout and hyperuricemia (serum uric acid > 7.0 mg/dl in men and >6.0 mg/dl in women) requiring uric acid lowering therapy.
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Febuxostat — One 40 mg tablet once a day for 6 months
  Other Names: Uloric

SUMMARY:
This study is being done to evaluate whether the medication, febuxostat, can improve the degree of insulin resistance and other features of the metabolic syndrome (high blood pressure, elevated insulin levels, excess body fat around the waist, and/or high cholesterol) by lowering uric acid levels in the blood.

DETAILED DESCRIPTION:
The metabolic syndrome (MS) is characterized by a constellation of metabolic features including dyslipidemia, hyperglycemia, hypertension, obesity, and insulin resistance. This cluster of features is strongly associated with type 2 diabetes, atherosclerotic cardiovascular disease, and increased cardiovascular and all-cause mortality. Hyperuricemia (elevated serum uric acid) is associated with insulin resistance and features of the MS in cross-sectional epidemiological studies. However, it remains unclear whether this association is causal or simply coincidental. If hyperuricemia CAUSES insulin resistance, then lowering serum uric acid by pharmacological means may result in improved insulin sensitivity and reversal of features of the metabolic syndrome. In some recent small studies, lowering serum uric acid with allopurinol was associated with improvement in some of the features and/or complications of the MS: Allopurinol use resulted in reduction in blood pressure in adolescents and improvement in exercise capacity in patients with chronic stable angina. A low urine pH is strongly associated with insulin resistance, and individual features of the metabolic syndrome. Similarly, a low fractional excretion of uric acid is also associated with metabolic syndrome feature. We therefore would like to examine the effect on febuxostat on these two parameters which have been linked with the metabolic syndrome.

The goal of this study is to evaluate whether pharmacological lowering of serum uric acid with the medication febuxostat is associated with improvement in the degree of insulin resistance and various features of the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Gout
* Hyperuricemia (serum uric acid > 7.0 mg/dl in men and >6.0 mg/dl in women).

Exclusion Criteria:

* Current treatment with insulin, azathioprine, mercaptopurine, or theophylline.
* Treatment with febuxostat, allopurinol or other uricosuric agents (including losartan, probenecid) within the past year
* Uncontrolled hypertension (clinic systolic blood pressure > 160 mmHg or diastolic blood pressure > 90 mmHg within the past 6 months)
* Uncontrolled diabetes mellitus (HbA1c > 7%)
* estimated GFR < 60 ml/min by MDRD
* Elevated liver function tests (AST or ALT greater than 3 times the upper limit of normal)
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naim M Maalouf, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marin M, Maalouf NM. Effects of pharmacological reversal of hyperuricemia on features of the metabolic syndrome in patients with gouty arthritis. J Investig Med. 2018 Oct;66(7):1031-1036. doi: 10.1136/jim-2018-000728. Epub 2018 Apr 4. PMID 29622755

RESULTS

PARTICIPANT FLOW:
Groups:
- Gout and Hyperuricemia: Adult patients (age > 21 years) with gout and hyperuricemia (serum uric acid > 7.0 mg/dl in men and >6.0 mg/dl in women) requiring uric acid lowering therapy.
  Febuxostat: One 40 mg tablet once a day for 6 months
Period: Overall Study
Arm/Group | Gout and Hyperuricemia
Started | 24
Visit 2 (2 Months) | 19
Visit 3 (4 Months) | 18
Visit 4 (6months) | 18
Completed | 18
Not Completed | 6
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: BMI
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
kg/m^2 | 33.4 (5.9)

2. Primary Outcome: Serum Uric Acid
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
mg/dl | 4.4 (1.1)

3. Primary Outcome: Serum Creatinine
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
mg/dl | 0.98 (0.22)

4. Primary Outcome: Ambulatory Systolic Blood Pressure
Description: Systolic BP by ambulatory blood pressure monitor.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
mmHg | 126 (14)

5. Primary Outcome: Ambulatory Diastolic Blood Pressure
Description: Diastolic BP by ambulatory blood pressure monitor.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
mmHg | 75 (9)

6. Primary Outcome: Serum Glucose
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
mg/dl | 107 (30)

7. Primary Outcome: Serum Insulin
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
mU/L | 14 (6.1)

8. Primary Outcome: Insulin Sensitivity Measured by HOMA (HOmeostasis Model Assessment)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Homeostatic model assessment for Insulin
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
Homeostatic model assessment for Insulin | 1.86 (.83)
Statistical Analysis 1: Comparison: Gout and Hyperuricemia; Test type: Superiority or Other; p = 0.66, t-test, 2 sided

9. Primary Outcome: Seum Total Cholesterol
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
mg/dl | 196 (46)

10. Primary Outcome: Serum HDL-cholesterol
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
mg/dl | 49 (16)

11. Primary Outcome: Serum Triglycerides
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
mg/dl | 175 (107)

12. Primary Outcome: Urine Uric Acid
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
mg/dl | 208 (137)

13. Primary Outcome: Urine Creatinine
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
mg/dl | 1332 (669)

14. Primary Outcome: Fractional Excretion UA
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % of serum uric acid excreted in urine
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
% of serum uric acid excreted in urine | 0.04 (0.02)

15. Primary Outcome: Urine pH
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Gout and Hyperuricemia
Number analyzed (Participants) | 18
pH | 5.58 (0.43)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Gout and Hyperuricemia
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gout and Hyperuricemia (N=24)
Abnormal Liver Function Test (Hepatobiliary disorders) | 0 (0) — Serum Liver function tests at months 2, 4 and 6.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes